CLINICAL TRIAL: NCT06387485
Title: A Study to Evaluate the Utilization of 3D Printed Models in Pre-Operative Planning
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ricoh USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SR-001
Record Dates: First submitted 2024-04-18; First posted 2024-04-29 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Sarcoma, Ewing; Chondrosarcoma; Osteosarcoma; Fibrous Histiocytoma; Fibrosarcoma
Keywords: bony tumor
MeSH Terms: conditions — Sarcoma, Ewing; Chondrosarcoma; Osteosarcoma; Histiocytoma, Benign Fibrous; Fibrosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard Imaging (Active Comparator): Participants in this arm will undergo tumor excision with prior planning utilizing only Imaging (CT or MRI) without development of a 3D printed model
  Interventions: Diagnostic Test: CT/MRI
- 3D Printed Anatomic Model (Experimental): Participants in this arm will have tumors excised with prior planning utilizing 3D printed models and Imaging (CT or MRI).
  Interventions: Device: 3D Printed Anatomic Model; Diagnostic Test: CT/MRI

INTERVENTIONS:
Device: 3D Printed Anatomic Model — Patient-specific 3D printed anatomic model for pre-surgical planning
  Arms: 3D Printed Anatomic Model
Diagnostic Test: CT/MRI — Standard imaging type for bony tumors

SUMMARY:
This prospective, multi-center, randomized controlled study aims to assess the efficacy of utilizing 3D printed models in preoperative planning for the excision of tumors involving bony structures within the body. The study is expected to last approximately 12 months and involve up to 150 subjects across up to 5 sites. Subjects will be randomized in a 1:1 ratio into either the experimental arm, utilizing 3D printed models and imaging, or the active comparator arm, using only imaging.

Primary endpoint: Operative time of surgical procedure.

Secondary endpoints: Reduction of blood loss, proportion of postoperative adverse events, and negative tumor margins.

Exploratory endpoints: Surgical planning ease, changes in surgical plan, and surgeon satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at least 13 years of age.
2. Subjects must have the ability to provide written informed consent.
3. Subjects must have tumor(s) invading bone and requiring surgical excision including but not limited to craniomaxillofacial, spine, long bone, and pelvis.
4. Subjects must be willing to have quality cross-sectional imaging that will allow for use to develop a 3D printed model.

Exclusion Criteria:

1. Pregnant or nursing women.
2. Subjects that have a serious systemic pathology.
3. Subjects that have clotting disorders.
4. Subjects that have uncontrolled hypertension.
5. Subjects that are HIV-positive.
6. Subjects that are unable to be randomized; i.e surgical team prefers to use either 3D model or standard cross-sectional imaging for surgical pre-planning.
7. Subject anatomy has changed substantially since the date medical imaging from which the model is derived was obtained (as applicable).
8. Subject is a poor surgical or poor study candidate which may include, any medical, social or psychological problem that could complicate the procedure.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Operative time | Incision to closure
  Operative time of surgical procedure based on incision and closure time

SECONDARY OUTCOMES:
Blood loss | Incision to closure
  Change in blood loss as determined by estimated blood loss and units of blood transfused (or blood products used) in mL.
Adverse Events | Surgery to 90 days post-surgery
  The proportion of ER visits and post operative procedure related adverse events/complications as reported at the 90-day Follow-Up Chart Review.
Tumor margin status | Post-surgery (+3 days)
  The proportion of negative tumor margins as determined by laboratory analysis.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Kaiser Permanente Oakland Medical Center, Oakland, California
  - William Beaumont University Hospital, Royal Oak, Michigan
  - The Ohio State University Wexner Medical Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No